CLINICAL TRIAL: NCT06236477
Title: Decreasing Emergence Delirium With Personalized Music
Acronym: DEAP Music
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Society for Pediatric Anesthesia (Other)
Responsible Party: Principal Investigator, Benjamin A Sanofsky, Anesthesiologist, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202309122
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Emergence Delirium
Keywords: Anesthesia; Music; Pediatric Anesthesia; Emergence Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Intervention Model Description: 1:1 parallel-group, superiority randomized controlled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized Music Group (Active Comparator): Those assigned to receive music will be asked to provide a short list of 5-10 songs familiar/well-known to the patient (specifically the song title and artist for each song). Songs will be downloaded onto an electronic mp3 player by the research staff member. The mp3 player will then be provided along with a portable Bluetooth speaker for use during the patient's perioperative period, loaded with the songs of their choice.
  Interventions: Behavioral: Personalized Music
- No Music Group (Placebo Comparator): Those not assigned to the personalized music group will receive standard care without music.
  Interventions: Behavioral: No Music

INTERVENTIONS:
Behavioral: Personalized Music — Music that is familiar to the child will be played via bluetooth speaker throughout their immediate perioperative care
  Arms: Personalized Music Group
Behavioral: No Music — Participants will receive standard care without music.
  Arms: No Music Group

SUMMARY:
This is a prospective randomized controlled trial in children 3-9 years of age undergoing myringotomies at Washington University in St. Louis to assess the impact of perioperative personalized music on the incidence of emergence agitation.

DETAILED DESCRIPTION:
Aim 1: Determine the efficacy of personalized music in decreasing the incidence of emergence agitation in pediatric patients undergoing myringotomies. Patients undergoing myringotomy procedures will be randomized to receive either standard care or personalized music during the perioperative period. The incidence of emergence agitation will be determined using the Pediatric Anesthesia Emergence Delirium scale.

Aim 2: Determine the efficacy of personalized music in reducing preoperative anxiety, postoperative pain, and maladaptive behavioral changes in pediatric patients following myringotomy procedures. Anxiety will be assessed in the preoperative holding area using the modified Yale Preoperative Anxiety Scale and the Induction Compliance Checklist (mask acceptance). Postoperative pain will be assessed in the post-anesthesia care unit using the Face, Legs, Activity, Cry, Consolability and Wong-Baker FACES scales. Behavioral changes will be measured using the Post Hospitalization Behavior Questionnaire via telephone calls on postoperative days 1 and 14 after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 3-9 years
* Presenting for unilateral or bilateral myringotomy under GA

Exclusion Criteria:

* Combined procedures
* Lack of interest in music (e.g., child who does not have musical preferences)
* Inability to hear music (patients with mild-moderate hearing loss who can perceive music will be included)
* Parent/guardian or patient refusal

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2026-03-28 (Estimated)

PRIMARY OUTCOMES:
Pediatric Anesthesia Emergence Delirium Scale | day of surgery
  Assessment scale for emergence delirium.Range 0-20, higher score indicates a worse outcome

SECONDARY OUTCOMES:
The modified Yale Preoperative Anxiety Scale | day of surgery
  Assessment scale for preoperative anxiety. Raw score 5-22; adjusted score range 23.33-100; higher scores indicates a worse outcome
Wong-Baker Faces Pain Rating Scale | day of surgery
  Pain scale. Range 0-10, higher score indicates a worse outcome
Face, Legs, Activity, Cry, Consolability scale | day of surgery
  Pain scale. Range 0-10, higher score indicates a worse outcome
Induction Compliance Checklist | day of surgery
  Assessment scale for anxiety during mask induction of anesthesia. Range 0-10, higher score indicates a worse outcome
Satisfaction survey | day of surgery
  Survey of parental satisfaction with perioperative care. A qualitative survey with discrete questions that contain "yes" or "no" or likert-style ratings ranging from "strongly disagree" to "strongly agree."
Post Hospitalization Behavior Questionnaire | 1 year
  Parental assessment of behavioral changes following surgery. Range 27-135, higher score indicates a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No